CLINICAL TRIAL: NCT00151112
Title: Comparison of Two Different Procedures for Plexus Anesthesia: Standard Position Versus Combination of Lateral Position and 20° Trendelenburg Position
Brief Title: Comparison of Two Different Procedures for Plexus Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principle Investigator: T. Weber, MD, Department of Anesthesiology and Intensive Care, University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01-Anast-05
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2008-09-11 (Estimated); Status verified 2008-09

CONDITIONS: Wounds and Injuries
Keywords: nerve block; regional anesthesia; injuries; diverse malformations
MeSH Terms: conditions — Wounds and Injuries | interventions — Patient Positioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): combination of lateral position and 20° Trendelenburg Position
  Interventions: Procedure: Positioning and plexus anesthesia
- 2 (Active Comparator): standard positioning
  Interventions: Procedure: Positioning and plexus anesthesia

INTERVENTIONS:
Procedure: Positioning and plexus anesthesia — positioning during plexus anesthesia

SUMMARY:
The purpose of this study is to investigate the influence of difference positioning on extension and efficacy of brachial plexus anesthesia at 20 minutes by using the axillary plexus block with supine positioning and a lateral positioning onto the non-anaesthetized side, combined with 20° Trendelenburg positioning.

ELIGIBILITY:
Inclusion Criteria:

* Single shot axillary block

Exclusion Criteria:

* Lateral position not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Extent of anesthesia | 20 minutes after acillary plexus block
Efficacy of anesthesia | 20 minutes after axillary plexus block

SECONDARY OUTCOMES:
Rate of failure | 20 minutes after axillary plexus block

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Weber, MD, Principal Investigator — Department of Anesthesiology and Intensive Care, University Hospital Münster
Locations (2):
- Germany (2):
  - BG Unfallklinik Murnau; Department of Anesthesiology, Murnau am Staffelsee
  - Department of Anesthesiology and Intensive Care, University Hospital Münster, Münster

REFERENCES:
- [Background] Bullmann V, Waurick R, Rodl R, Hulskamp G, Orlowski O, van Aken H, Winkelmann W, Weber TP. [Corrective osteotomy of the humerus using perivascular axillary anesthesia according to Weber in a patient suffering from McCune-Albright syndrome]. Anaesthesist. 2005 Sep;54(9):889-94. doi: 10.1007/s00101-005-0874-6. German. PMID 15947897